CLINICAL TRIAL: NCT03855631
Title: Exploiting Epigenome Editing in Kabuki Syndrome: a New Route Towards Gene Therapy for Rare Genetic Disorders
Acronym: Epi-KAB
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Association Française contre les Myopathies Telethon (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0242
Record Dates: First submitted 2019-02-22; First posted 2019-02-27 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Kabuki Syndrome 1
Keywords: Kabuki syndrome CRIPSR/Cas9 KMT2D
MeSH Terms: conditions — Kabuki syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin fibroblast from 4 KS patients with KMT2D mutation and sex matched parents
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kabuki syndrome/ unaffected parents: Intervention on primary cultured cells from 4 patients with KS and sex match parents
  Interventions: Genetic: Intervention on primary cultured cells

INTERVENTIONS:
Genetic: Intervention on primary cultured cells — The intervention includes primary cultured cells, reprograming them into mesenchymal stem cells and CRISPR/Case9 gene therapy treatment on patients' cells

SUMMARY:
Starting from isolating primary cells from affected patients, an in vitro disease model system for KS will be developed. Using alternative strategies to obtain patient-derived mesenchymal stem cells, an integrative approach will be adopted for defining both the transcriptional and epigenetic regulatory networks perturbed upon the loss of function of KMT2D. Combining the self-renewal potential of mesenchymal stem cells (MSCs) with CRISPR/Cas9 technology, an epigenome editing approach as therapeutic strategy to rescue the activity of MLL4 will be developed.

A step forward is expected towards the understanding of those the molecular mechanisms governing the aetiology of Kabuki Syndrome (KS) and that the proposed in vitro disease model will provide to the scientific community an experimental system to study the KS. Importantly, the aim is to define the molecular bases of KS and to develop a therapeutic strategy that could ameliorate some of the abnormalities associated with KS.

DETAILED DESCRIPTION:
Main and secondary objectives :

The main objective is to study the pathological role of ML mutations in KS to facilitate the identification and characterization of therapeutic strategies to improve the symptoms of patients with KS. Due to the lack of treatment in the KS, the aim is to develop a model of this disease from fibroblasts from patients and reprogram them into mesenchymal stem cells. This approach will generate a KS-specific stem cell bio-bank, allowing the identification of common disturbances caused by the loss of function (LoF) of KMT2D. The impact of the KMT2D LoF on transcription but also the epigenetic mechanisms activated during MSC differentiation will be described. Finally, the therapeutic potential of an epigenome "editing" approach to increase the expression of the wild KMT2D allele to restore the functional activity of MLL4 in treated MSCs will be evaluated.

The secondary objective is to evaluate the ability to return to normal after CRISPR/Case9 gene therapy treatment on patients' cells

Methodology (design study, population, description of groups (if applicable), inclusion criteria, non-inclusion, main and secondary judgment criteria, number of subjects to be included, statistical analysis...) :

Starting from primary cells isolated from affected patients, an in vitro model of the disease will be developed. An integrative but alternative strategy approach to obtain mesenchymal stem cells derived from patients to define normal and abnormal transcription and epigenetic circuits during KMT2D LoF will be adopted. By combining the autonomous renewal potential of MSCs with CRISPR/Cas9 technology, an approach to "editing" the epigenome for therapeutic purposes to restore MLL4 activity will be developed.

This project will represent a step forward in understanding the molecular mechanisms responsible for KS. The in vitro model will provide the scientific community with an experimental system to study KS. Finally, the aim is to define the molecular basis of KS and develop a therapeutic strategy to improve certain symptoms in patients with KS.

Process (number of visits, duration of inclusions, duration of follow-up):

8 people will be included: 4 patients with Kabuki syndrome authenticated by the molecular genetics study of the KMT2D gene.

4 parents of the same sex as the patient

Feasibility :

In the clinical genetics department of the Montpellier University Hospital, more than 40 patients with Kabuki syndrome are followed.

Impacts / prospects :

The identification of the consequences of mutations in the KMT2D gene on epigenetic mark changes and cellular structural changes as well as the attempt at gene correction by CRISPR/Cas9 will provide a better understanding of the disease (and the genes that are deregulated by post-KMT2D epigenetic changes) and will also open a promising path for gene therapy by CRISPR/Cas9 method.

ELIGIBILITY:
Inclusion Criteria:

1. For the patient = to have a Kabuki syndrome authenticated by molecular genetics (proof of mutation in the KMT2D gene)
2. For parents = having the same sex as your child
3. To be affiliated to a French social security system
4. Authorize the participation of the study

Exclusion Criteria:

1. Not be affiliated to a social security scheme (CMU is included)
2. Existence of a significant coagulation ruble (especially thrombocytopenic purpura in Kabuki patients with platelet counts < 20,000 Units).
3. Genetic skin disease responsible for poor healing
4. Refusal to participate in the child's and/or parent's study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric population with KS and healthy adult (unaffected sex match parents of patients)
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
success rate of fibroblasts culture | one year maximum after inclusion
  The aim is to establish a model of KS disease from fibroblasts from patients

SECONDARY OUTCOMES:
success rate of turning fibroblasts into mesenchymal stem cells | one year maximum after inclusion
  The aim is to determine the success rate of turning fibroblasts into mesenchymal stem cells
success rate of CRISPR/Case9 gene therapy treatment on patients' cells | one year maximum after inclusion
  The aim is to evaluate the ability to return to normal after CRISPR/Case9 gene therapy treatment on patients' cells

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Zippo, PhD, Principal Investigator — Center of Integrative Biology
Locations (1):
- Arnaud de villeneuve Hospital, Montpellier, Herault, France